CLINICAL TRIAL: NCT00378846
Title: A Study Evaluating the Agreement of Devices for Measuring Temperature in Children
Brief Title: Three Different Types of Thermometers in Measuring Temperature in Young Patients With Fever and Without Fever
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: 060118; 06-C-0118; NCI-P6842; CDR0000496917
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Fever, Sweats, and Hot Flashes
Keywords: fever, sweats, and hot flashes
MeSH Terms: conditions — Fever; Hot Flashes

INTERVENTIONS:
Procedure: infrared thermography

SUMMARY:
RATIONALE: Comparing results of three different thermometers used to measure body temperature may help doctors find the most accurate thermometer to detect fever and plan the best treatment.

PURPOSE: This clinical trial is studying three different types of thermometers to measure temperature in young patients with fever and without fever.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine agreement between three different types of temperature-measuring instruments: the temporal artery scanner, the digital oral thermometer, and the infrared tympanic thermometer calibrated to an oral setting, in pediatric patients who are febrile and afebrile.

Secondary

* Determine similarities or differences in the percent of fevers detected with oral, ear, and temporal artery monitoring in these pediatric patients.
* Determine differences in agreement of the various temperature devices in non-neutropenic pediatric patients versus neutropenic pediatric patients.

OUTLINE: This is a prospective study.

During an afebrile episode, the patient's temperature is measured twice using the following 3 devices: a temporal artery scanner, a digital oral thermometer, and an infrared tympanic thermometer calibrated to an oral setting (total of 6 temperature measurements per afebrile episode).

During a febrile episode, the patient's temperature is measured twice using all 3 devices as above, and then at 2 and 4 hours after administration of an antipyretic medication (total of 18 temperatures per febrile episode).

Patients' temperatures are recorded for a maximum of 3 afebrile or febrile episodes.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Febrile or afebrile
* Patient at the Mark O. Harfield Clinical Research Center

  * Previously enrolled in an IRB-approved Clinical Center protocol

PATIENT CHARACTERISTICS:

* Able to hold an oral thermometer in mouth
* No acute life-threatening infection
* No ear, nose, or throat (aural) abnormalities
* No severe mucositis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent enrollment on a behavioral research study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2006-03; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Agreement between the temporal artery scanner, digital oral thermometer, and infrared tympanic thermometer calibrated to an oral setting in pediatric patients who are febrile and afebrile

SECONDARY OUTCOMES:
Similarities or differences in the percent of fevers detected with oral, ear, and temporal artery monitoring
Differences in agreement of the various temperature devices

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Walsh, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States